CLINICAL TRIAL: NCT00704028
Title: A Multi-Center, Randomized, Controlled Study to Investigate the Safety and Tolerability of Intravenous Ferric Carboxymaltose (FCM) vs. Iron Dextran in Treating Iron Deficiency Anemia
Brief Title: Safety and Tolerability of Ferric Carboxymaltose (FCM) Versus Iron Dextran in Treating Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT08020
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): 15 mg/kg up to a maximum of 750 mg at 100 mg per minute weekly to a maximum cumulative dose of 2,250 mg.
  Interventions: Drug: Ferric Carboxymaltose
- Iron Dextran (Active Comparator): As determined by the investigator to a maximum cumulative dose of 2,250 mg.
  Interventions: Drug: Iron Dextran

INTERVENTIONS:
Drug: Ferric Carboxymaltose — 15 mg/kg up to a maximum of 750 mg at 100 mg per minute weekly to a maximum cumulative dose of 2,250 mg.
  Arms: Ferric Carboxymaltose (FCM)
Drug: Iron Dextran — As determined by the investigator to a maximum cumulative dose of 2,250 mg.
  Other Names: Dexferrum, INFeD
  Arms: Iron Dextran

SUMMARY:
The objective of this study is to evaluate the safety of FCM in patients with anemia who are not dialysis dependent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age and able to give informed consent
* Iron deficiency is the primary etiology of anemia
* History of intolerance or an unsatisfactory response to oral iron
* Screening Visit central laboratory Hgb ≤11 g/dL
* Screening Visit ferritin ≤100 ng/mL or ≤300 when TSAT was ≤30%

Exclusion Criteria:

* Previous participation in a FCM trial
* Known hypersensitivity reaction to FCM or iron dextran
* Requires dialysis for treatment of chronic kidney disease
* Current anemia not attributed to iron deficiency
* Received IV iron, RBC transfusion(s), or antibiotics 10 days prior and during the screening phase
* Anticipated need for surgery during the 30 day period prior to screening or during the study period
* AST or ALT greater than 1.5 times the upper limit of normal
* Received an investigational drug within 30 days of screening
* Women who are breastfeeding
* Pregnant or sexually-active females who are not willing to use an effective form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Pre-assignment Details: One subject randomized to iron dextran never received study drug and was discontinued due to subject request.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran
Started | 82 | 78 (A subject randomized to iron dextran never received study drug and was d/c due to subject request.)
Completed | 70 | 57
Not Completed | 12 | 21

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran | Total
Number analyzed (Participants) | 82 | 78 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 72 | 62 | 134
  >=65 years | 10 | 15 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.64) | 48.2 (17.10) | 47.2 (15.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 69 | 142
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 82 | 78 | 160

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Reported Treatment-emergent Adverse Events (AE's)
Time Frame: Day 0 through end of study (Day 42), or 28 days after the last dose of study drug whichever was longer
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran
Number analyzed (Participants) | 82 | 78
participants | 60 | 59

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ferric Carboxymaltose (FCM) | Iron Dextran
Serious Adverse Events (participants affected / at risk) | 5/82 | 3/78
Other Adverse Events (participants affected / at risk) | 45/82 | 54/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=82) | Iron Dextran (N=78)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=82) | Iron Dextran (N=78)
Diarrhea (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 5 | 4
Hypersensitivity (Immune system disorders) | 0 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 0
Dizziness (Nervous system disorders) | 6 | 4
Headache (Nervous system disorders) | 6 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less